CLINICAL TRIAL: NCT01033448
Title: An Open-Label, Multi-Center Study Evaluating the Effect on Viral Activity and the Safety and Tolerability of Extended Treatment of Pegasys® (Peginterferon Alfa 2a ) in Combination With Copegus® (Ribavirin) in Genotype 1, 2 and 3 Chronic Hepatitis C Patients Defined as Slow Responders/Non-RVR
Brief Title: A Study of Extended Therapy of PEGASYS (Peginterferon Alfa-2a) in Combination With COPEGUS (Ribavirin) in Patients With Chronic Hepatitis C and Slow Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21778
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: COPEGUS; Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: COPEGUS — COPEGUS 800 mg or 1000-1200 mg po for 24 weeks
Drug: peginterferon alfa-2a [Pegasys] — PEGASYS 180 micrograms sc once weekly for 24 weeks

SUMMARY:
This open-label, multi-center study will evaluate the safety and tolerability and the effect on viral activity of a combined PEGASYS and COPEGUS extended therapy in patients with chronic hepatitis C with genotype 1, 2 and 3. Patients who completed 48 weeks (genotype 1) or 24 weeks (genotype 2 and 3) of standard treatment with PEGASYS and COPEGUS and were identified as slow virological responders will be enrolled in this study in order to receive additional 24 weeks of treatment. PEGASYS 180 micrograms will be administered sc once weekly and COPEGUS will be administered as 800 mg, or 1000-1200 mg daily oral doses. The anticipated time on study treatment is 24 weeks. The target sample size is 50-150 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >/= 18 years of age
* Chronic hepatitis C, genotype 1, 2, 3
* Compensated liver disease
* Patients who completed 48 weeks or 24 weeks of standard treatment with PEGASYS and COPEGUS and were identified as slow virological responders

Exclusion Criteria:

* Decompensated liver disease
* Signs or symptoms of hepatocellular carcinoma
* Uncontrolled hypoglycaemia, hyperglycaemia and diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- Israel (20):
  - Haemek Hospital; Gastroenterology, Afula
  - Clalit City Ashdod MC; Liver Clinic, Ashdod
  - Batyamon; Liver Unit, Bat Yam
  - Soroka Medical Center; Gastroenterology, Beersheba
  - Rambam Medical Center; Gastroenterology - Liver Unit, Haifa
  - Bnei-Zion Medical Center; Gastroenterology, Haifa
  - Carmel Hospital; Liver Unit, Haifa
  - Wolfson Hospital; Gastroenterology Unit, Holon
  - Hadassah Hospital; Liver Unit, Jerusalem
  - Clalit Strauss MC, Jerusalem
  - Meir Medical Center; Gastroenterology, Kfar Saba
  - Naharyia / Western Galilee MC; Gastro Unit, Nahariya
  - Holy Family Medical Center; Gastroenterology, Nazareth
  - Rabin Medical Center; Gastroenterology - Liver Unit, Petah Tikva
  - Kaplan Medical Center; Gastroenterology Unit, Rehovot
  - Clalit Pinsker Rishon; Liver Clinic, Rishon LeZiyyon
  - Rebecca Sieff Medical Center; Liver Unit, Safed
  - Maccabi Health Services MC, Tel Aviv
  - Poria Hospital; Gastroenterology, Tiberias
  - Assaf Harofeh; Gastroenterology, Ẕerifin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from Study NCT01429792 with genotype 1 Chronic Hepatitis C (CHC) and were 'Slow Responders' were eligible to enroll in this treatment extension study. Participants from Study NCT01429792 with genotype 2 and 3 CHC and were non-Rapid Virologic Response (RVR) were eligible to enroll in this treatment extension study.
Pre-assignment Details: A total of 59 participants were enrolled in the study and 47 of them completed the study.
Groups:
- Pegylated Interferon (Peginterferon) Alfa-2a: Participants received pegylated interferon alfa-2a 180 microgram (mcg) in 0.5 milliliter (mL) solution administered subcutaneous (SC) once weekly for 24 weeks. Ribavirin was administered for 24 weeks
Period: Overall Study
Arm/Group | Pegylated Interferon (Peginterferon) Alfa-2a
Started | 59
Completed | 47
Not Completed | 12
Not completed — Withdrawal by Subject | 4
Not completed — Positive HCV-RNA at week 48 | 1
Not completed — Lost to Follow-up | 3
Not completed — Withdrew due to other reasons | 3
Not completed — Unknown disposition | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants were included in the baseline population.
Arm/Group | Pegylated Interferon (Peginterferon) Alfa-2a
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: End of Treatment Response Rate at Week 72 in Genotype 1
Description: End of treatment response rate at Week 72 was reported for genotype 1.
Time Frame: Week 72
Population: Participants with genotype 1 CHC at Week 72.
Measure: Number; unit: Percentage of Participants
Groups:
- CHC Genotype 1: Participants received pegylated interferon alfa2a 180 microgram (mcg) in 0.5 milliliter (mL) solution administered subcutaneous (SC) once weekly for 24 weeks. Ribavirin was administered 1000-1200 mg ribavirin were administered orally in split doses in the morning and in the evening for 24 weeks.
Arm/Group | CHC Genotype 1
Number analyzed (Participants) | 44
Percentage of Participants | 68.2

2. Primary Outcome: End of Treatment Response in Genotype 2 and 3
Description: End of treatment response rate at Week 48 was reported for genotype 2 and 3.
Time Frame: Week 48
Population: Participants with CHC Genotype 2 and 3 at Week 48.
Measure: Number; unit: Percentage of Participants
Groups:
- CHC Genotype 2 and 3: Participants received peginterferon alfa-2a 180 mcg in 0.5 mL solution administered SC once weekly plus ribavirin 800 mg orally in split doses in the morning and in the evening for 24 weeks.
Arm/Group | CHC Genotype 2 and 3
Number analyzed (Participants) | 15
Percentage of Participants | 66.7

3. Primary Outcome: Sustained Viral Response (SVR) Rates in CHC Genotype 1
Description: Sustained Viral Response, undetectable HCV-RNA 24 weeks after the end of treatment for genotype 1.
Time Frame: Week 96
Population: Participants with CHC genotype 1 at Week 96
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CHC Genotype 1
Number analyzed (Participants) | 44
Percentage of participants | 46.5 [31.2 to 62.3]

4. Primary Outcome: SVR Rates in Genotype 2 and 3.
Description: Sustained Viral Response, undetectable HCV-RNA 24 weeks after the end of treatment for genotype 2 and 3.
Time Frame: Week 72
Population: Participants with CHC Genotype 2 & 3 at week 72.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CHC Genotype 2 and 3
Number analyzed (Participants) | 15
Percentage of participants | 60.0 [32.3 to 83.7]

5. Secondary Outcome: Percentage of Participants With Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Week 96
Population: All enrolled participants were analyzed
Measure: Number; unit: Percentage of Participants
Groups:
- Pegylated Interferon (Peginterferon) Alfa2a: Participants received pegylated interferon alfa2a 180 microgram (mcg) in 0.5 milliliter (mL) solution administered subcutaneous (SC) once weekly for 24 weeks. Ribavirin was administered for 24 weeks.
Arm/Group | Pegylated Interferon (Peginterferon) Alfa2a
Number analyzed (Participants) | 59
Percentage of Participants | 40.7

ADVERSE EVENTS:
Time Frame: Baseline to Week 96
Description: Safety population included all enrolled participants.
Groups:
- Pegylated Interferon Alfa2a (Peginterferon): Participants received pegylated interferon alfa2a 180 microgram (mcg) in 0.5 milliliter (mL) solution administered subcutaneous (SC) once weekly for 24 weeks. Ribavirin was administered for 24 weeks.
Arm/Group | Pegylated Interferon Alfa2a (Peginterferon)
Serious Adverse Events (participants affected / at risk) | 5/59
Other Adverse Events (participants affected / at risk) | 14/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated Interferon Alfa2a (Peginterferon) (N=59)
Pyrexia (General disorders) | 1
Anal Abscess (Infections and infestations) | 1
Anaesthesia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Pregnancy of partner (Social circumstances) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated Interferon Alfa2a (Peginterferon) (N=59)
Anaemia (Blood and lymphatic system disorders) | 12
Neutropenia (Blood and lymphatic system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.